CLINICAL TRIAL: NCT01282398
Title: Prevention of Progression of Portal Hypertension in Compensated Cirrhosis Using Selective Hepatic Vasodilators. A Double-blind, Multicenter,Randomized Controlled Trial
Brief Title: Study About Simvastatin in Portal Hypertension in Compensated Cirrhosis
Acronym: SIMPRO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Candido Villanueva, Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IIBSP-SIM-2010-06
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Portal Hypertension.; Liver Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- simvastatin (Experimental): The experimental group will take simvastatin 40mg for at least two years.
  Interventions: Drug: Simvastatin
- placebo (Placebo Comparator): the control group wiil take placebo pills for at least two years.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Simvastatin — The experimental group will take 40 mg each 24 hours for at least two years.
  Arms: simvastatin
Drug: placebo — the control group wiil take placebo pills for at least two years.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether simvastatin is effective in the prevention of progression of porta hypertension in compensated cirrhosis patients.

DETAILED DESCRIPTION:
Decompensation of cirrhosis is associated with a dramatic reduction of survival. Progression of portal hypertension (PHT) is the main determinant of decompensation that appears when portal pressure gradient (PPG) is ≥10mmHg (clinically significant HTP). 40% of compensated cirrhotic patients have mild PHT. However, with progression of disease 41% develop clinically significant PHT. In cirrhosis, PHT results from increased resistance to blood flow, with a dynamic component due to decreased nitric oxide (NO) bioavailability. In advanced disease increased portal venous inflow also contributes to PHT. Beta-blockers have not been useful in compensated cirrhosis with mild PHT. In early cirrhosis, vasodilators may be more adequate. Statins, drugs that inhibit the activity of HMG-CoA reductase, induce selective hepatic vasodilation due to an enhanced bioavailability of NO. Acutely, they decreases hepatic resistance, while with long-term use statins decreases PPG without deleterious effects on systemic circulation. This multicenter, randomized, double-blind placebo-controlled study is aimed at assessing whether treatment with simvastatin may prevent progression of mild PHT (with PPG between 6 and 10 mmHg) to clinically significant PHT. Patients with compensated cirrhosis, without previous decompensation, without esophageal varices at risk and with PPG between 6 and 10 mmHg will be included. The calculated sample size is 80 patients and the duration of the study 4 years (2 years including and a follow-up of at least 2 year).

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis diagnosed by previous biopsy or by clinical, laboratory, ultrasound
* Portal hypertension gradient between6 mmHg and10 mmHg
* Absence of esophageal and gastric varices or small esophageal varices without red signs
* Absence previous episodes of gastrointestinal hemorrhage, ascites, encephalopathy or jaundice
* Written informed consent

Exclusion Criteria:

* Age <18 and> 80 years,
* Presence or history of ascites, clinical or ultrasound,
* Previous decompensation of liver cirrhosis, ascites or SBP, bleeding varices, large varices, hepatic encephalopathy, jaundice,
* Thrombosis splenoportal,
* Hepatocellular carcinoma;
* Child-Pugh >7 point
* Any comorbidity that leads to a restriction therapy and / or a life expectancy <12 months
* Absolute contraindication to treatment with statins or allergy Simvastatin;
* Concomitant potent CYP3A4 inhibitors (eg., itraconazole, ketoconazole, protease inhibitors, HIV, erythromycin, clarithromycin, telithromycin and nefazodone),
* Pretreatment (<1 month) with simvastatin or other lipid-lowering,
* Previous episodes of rhabdomyolysis,
* Active alcoholic hepatitis,
* Refusal to participate in the study or the informed consent claim;
* Pre-treatment with beta blockers or nitrates, or endoscopic treatment for varicose veins or portosystemic derivations;
* Pregnancy and lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
the treatment of portal hypertension with simvastatin may prevent progression of portal hypertension | 4 years
  The main objective is to assess whether, in patients with compensated cirrhosis and mild portal hypertension (GPP between 6 and 10mmHg), the treatment of portal hypertension with simvastatin may prevent progression of portal hypertension and prevent the development of clinically significant HTP (defined GPP by a ≥ 10 mmHg)

SECONDARY OUTCOMES:
Portal hypertension complications | four years
  Development of complications related to portal hypertension (gastrointestinal bleeding related to portal hypertension, ascites, hepatic encephalopathy).
Adverse effects | four years

CONTACTS AND LOCATIONS:
Overall Officials: Candido Villanueva, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Abraldes JG, Albillos A, Banares R, Turnes J, Gonzalez R, Garcia-Pagan JC, Bosch J. Simvastatin lowers portal pressure in patients with cirrhosis and portal hypertension: a randomized controlled trial. Gastroenterology. 2009 May;136(5):1651-8. doi: 10.1053/j.gastro.2009.01.043. Epub 2009 Jan 24. PMID 19208350
- [Result] Groszmann RJ, Garcia-Tsao G, Bosch J, Grace ND, Burroughs AK, Planas R, Escorsell A, Garcia-Pagan JC, Patch D, Matloff DS, Gao H, Makuch R; Portal Hypertension Collaborative Group. Beta-blockers to prevent gastroesophageal varices in patients with cirrhosis. N Engl J Med. 2005 Nov 24;353(21):2254-61. doi: 10.1056/NEJMoa044456. PMID 16306522
- [Result] Villanueva C, Aracil C, Colomo A, Hernandez-Gea V, Lopez-Balaguer JM, Alvarez-Urturi C, Torras X, Balanzo J, Guarner C. Acute hemodynamic response to beta-blockers and prediction of long-term outcome in primary prophylaxis of variceal bleeding. Gastroenterology. 2009 Jul;137(1):119-28. doi: 10.1053/j.gastro.2009.03.048. Epub 2009 Apr 1. PMID 19344721
- [Result] Zafra C, Abraldes JG, Turnes J, Berzigotti A, Fernandez M, Garca-Pagan JC, Rodes J, Bosch J. Simvastatin enhances hepatic nitric oxide production and decreases the hepatic vascular tone in patients with cirrhosis. Gastroenterology. 2004 Mar;126(3):749-55. doi: 10.1053/j.gastro.2003.12.007. PMID 14988829
- [Derived] Marrache MK, Rockey DC. Statins for treatment of chronic liver disease. Curr Opin Gastroenterol. 2021 May 1;37(3):200-207. doi: 10.1097/MOG.0000000000000716. PMID 33654016